CLINICAL TRIAL: NCT00924079
Title: Pharmacokinetic Study of Oral Nalbuphine in Normal Healthy Subjects
Brief Title: The Development of Oral Nalbuphine Dosage Form
Acronym: NAL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Ho Shung-Tai/Professor of the department of anesthsiology, Department of anesthsiology of Tri-service General Hospitial
Allocation: Non-Randomized | Model: Crossover | Masking: None
Other Study IDs: NAL001; TSGHIRB096-02-010-I
Record Dates: First submitted 2009-06-17; First posted 2009-06-18 (Estimated); Last update posted 2009-06-19 (Estimated); Status verified 2009-06

CONDITIONS: Healthy
Keywords: Analysis of plasma concentration of nalbuphine
MeSH Terms: interventions — Nalbuphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- nalbuphine (Experimental)
  Interventions: Drug: nalbuphine

INTERVENTIONS:
Drug: nalbuphine — oral dosage form, 66 mg, single dose

SUMMARY:
The purpose of this study is to investigate possible responses to pharmacokinetic properties for nalbuphine oral formulations in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Normal healthy adult subjects between 20-40 years of age.
* Body weight within 80-120% of ideal body weight. Ideal body weight = (height-80)0.7
* Acceptable medical history and physical examination including:

  * Normal chest X-ray and ECG results within six months prior to Period I dosing.
  * No particular clinical significance in general disease history within two months prior to Period I dosing.
* Acceptable clinical laboratory determinations without significant deviation from normal values within two months prior to Period I dosing, which includes:

  * AST (SGOT)
  * ALT (SGPT)
  * Gama-GT
  * alkaline phosphatase
  * total bilirubin
  * albumin
  * glucose
  * BUN
  * uric acid
  * creatinine
  * total cholesterol
  * triglyceride(TG)
* Acceptable hematology within two months prior to the study, which includes hemoglobin, hematocrit, red blood cells, MCV, MCH, MCHC, white blood cells, differential white blood cells and platelets.
* Acceptable urinalysis within two months prior to the study, which includes pH, blood, glucose and protein.
* Signed the written informed consent to participate in this study.

Exclusion Criteria:

* Recent history of drug or alcohol addiction or abuse.
* A clinically significant disorder involving the cardiovascular, respiratory, renal, gastrointestinal, immunologic, hematologic, endocrine or neurologic system(s) or psychiatric disease (as determined by the clinical investigator).
* History of allergic response(s) to nalbuphine or related drugs.
* History of clinically significant allergies including drug allergies or allergic bronchial asthma.
* Evidence of chronic or acute infectious diseases.
* Any clinically significant illness or surgery during the four weeks prior to Period I dosing (as determined by the clinical investigator).
* Taking any drug known to induce or inhibit hepatic drug metabolism within one month prior to the beginning of the study.
* Receiving any investigational drug within one month prior to Period I dosing.
* Taking any prescription medication or any nonprescription medication within two weeks prior to Period I doing.
* Donating greater than 150 ml of blood within two months prior to Period I dosing or donating plasma (e.g., plasmapheresis) within 14 days prior to Period I dosing. All subjects will be advised not to donate blood for four weeks after completing the study.
* Consumption of caffeine, xanthine-containing products (i.e., coffee, tea, caffeine-containing sodas, colas and chocolate, etc.) and/or alcohol at least 48 hours prior to days on which dosing is scheduled and during the periods when blood samples are being collected.
* Any other medical reason as determined by the clinical investigator.
* Patient is pregnant or breastfeeding. Women of childbearing potential must have a negative urine pregnancy test at Baseline.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-09; Primary Completion 2009-11 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic parameter eq Cmax, AUC, Cl, T1/2 | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Tri-Service General Hospitial, Taipei, Taiwan